CLINICAL TRIAL: NCT04536233
Title: The Safety and Effectiveness of Mesenchymal Stem Cell-derived Pleiotropic Factors on Wound Healing in Endonasal Surgeries
Brief Title: Effects of MSCs Derived Pleiotropic Factors on Wound Healing in Endonasal Surgeries
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHIN-PLAGH-MP-05
Record Dates: First submitted 2020-08-30; First posted 2020-09-02 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: MSCs Derived Pleiotropic Factors on Wound Healing in Endonasal Surgeries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator)
  Interventions: Other: physiological saline
- experimental group (Experimental)
  Interventions: Biological: MSCs Derived Pleiotropic Factors

INTERVENTIONS:
Biological: MSCs Derived Pleiotropic Factors — The pleiotropic factor derived from mesenchymal stem cells was injected on the wound
  Arms: experimental group
Other: physiological saline — The physiological saline was injected on the wound
  Arms: control group

SUMMARY:
Nasal trauma, deviated nasal septum, sinusitis, nasal polyps and other nasal benign diseases are common clinical diseases and require endoscopic sinus surgery. The proper application of the surgical procedure as well as ensuring high quality of wound healing, is also important to achieve successful results in endoscopic sinus surgery. If good quality wound healing cannot be achieved in the surgical field,synechiae and anatomic defects can occur that may require revision surgeries.

Mesenchymal stem cells play an active role in the treatment of many diseases. it primarily exerts therapeutic effects through paracrine. In this study, the effect of mesenchymal stem cell-derived multipotent factors on mucosal repair after nasal surgery was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 60 years old;
2. The clinical diagnosis is nasal trauma, nasal septum deviation, sinusitis, and nasal polyps requiring endoscopic surgery;
3. The patient's physical and mental state is stable, and he can return to the hospital regularly for follow-up examinations and cooperate to complete the experiment;

Exclusion Criteria:

1. Younger than 18 or older than 60;
2. Clinical diagnosis of nasal malignancies, or uncontrolled severe infectious diseases;
3. Past medical history of mental illness, malignant tumor, nose surgery;
4. People with serious underlying diseases (hypertension, diabetes, rheumatism, asthma) require long-term medication;
5. Long-term smoking, more than 5 cigarettes per day;
6. Work or daily life environment is exposed to large amounts of dust and chemical raw materials;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-10 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing evaluation | 2 months
  Lund-Kennedy scoring method；under video nasal endoscopy. Including five aspects of polyps, edema, rhinorrhea, scars, and scabs, each score is 0-2 points. Polyp: 0 points means no polyps, 1 point means polyps only in the middle nasal passage, 2 points means polyps beyond the middle nasal passage. Edema: 0 points means no edema, 1 point means mild edema, 2 points means severe edema. Rhinorrhea: 0 points means no rhinorrhea, 1 point means clear and thin nose, 2 points means rhinorrhea is sticky and purulent. Scar: 0 points means no scars, 1 points means mild scars, 2 points means severe scars. Scab formation: 0 points means no scab formation, 1 point means mild scab formation, and 2 points means severe scab formation. Each side 0-10 points, a total of 20 points, the lower the score indicates that the patient's symptoms are lighter.

IPD SHARING:
Plan to Share IPD: Undecided
If there are researchers who need relevant data, they can apply to us